CLINICAL TRIAL: NCT01625598
Title: A Multicenter Masked Study to Compare Analysis of the Detection Program IDx-DR Against Standard of Care Clinical Examination by Ophthalmologists to Differentiate Levels of Diabetic Retinopathy and Diabetic Macular Edema
Brief Title: Computer Detection of Diabetic Retinopathy Compared to Clinical Examination
Acronym: CDDR
Status: Completed | Type: Observational
Sponsor: Digital Diagnostics, Inc. (Industry)
Collaborators: University of Pennsylvania (Other); University of Iowa (Other); The University of Texas Health Science Center, Houston (Other); Iowa Eye Center, Cedar Rapids IA (Unknown); VitreoRetinal Surgery, PA (Other); Retina Consultants Houston (Other); Barnet Dulaney Perkins Eye Centers (Network)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2012-05-25; First posted 2012-06-21 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Retinopathy
Keywords: Nonproliferative diabetic retinopathy; diabetic macular edema; proliferative diabetic retinopathy; ophthalmologists; dilated eye exam
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- People with diabetes: People with diabetes who are referred to an ophthalmologist for a dilated eye examination
  Interventions: Procedure: Photography of the retina; Procedure: Retinal photography

INTERVENTIONS:
Procedure: Photography of the retina — Every subject will undergo photography of the retina in both eyes
Procedure: Retinal photography — Device
  Subjects will have photography of both eyes

SUMMARY:
The hypothesis is that computer detection of the severity of diabetic retinopathy including the presence of clinically significant macular edema is not inferior to the detection using a dilated eye examination by a Board-certified ophthalmologist.

DETAILED DESCRIPTION:
The project is a multicenter, observational study to compare the accuracy of the IDX-DR computer detection system to board certified ophthalmologists performing dilated eye examination at identifying between no or mild NPDR without clinically significant diabetic macular edema from more than mild NPDR with or without CSDME. Approximately 400-600 persons with diabetes will be recruited through 5 clinical centers. The ophthalmologist who examines the patient will evaluate and record the status of the eye based on his/her clinical examination. The study subjects will then have two fundus photographs taken of each eye. The photographic images will be transferred to a central Reading Center at the University of Pennsylvania and interpreted by professional graders. The Reading Center will then transfer the images to IDx-DR, the computer detection system. IDx-LLC, the Sponsor of this study, will have no access to the images. Data from the Reading Center interpretation will be considered the "gold standard". The results of the clinical examination and IDX-DR will be compared against this gold standard as well as against each other.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of diabetes mellitus
* subject understands study and has signed informed consent
* no history of any other retinal vascular disease, glaucoma, or other disease that may affect the appearance of the retina or optic disc (refractive error and ocular surface disease are allowed);
* other than cataract surgery, no history of intraocular surgery, ocular laser treatments for any retinal disease, or ocular injections for diabetic macular edema or proliferative disease
* no media opacity precluding good retinal photography
* age 18 or older

Exclusion Criteria:

* no diagnosis of diabetes mellitus
* potential subject cannot understand study or informed consent
* a history of retinal vascular disease other than due to diabetic retinopathy, glaucoma, or other disease that may affect the appearance of the retina or optic disc
* previous intraocular surgery other than cataract; previous laser to the retina; or previous intraocular injections for the treatment of diabetic retinopathy
* a media opacity in either eye that is severe enough to preclude good retinal photography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with diabetes, eighteen years of age or older, who have been referred to an ophthalmologists for a dilated eye examination to detect diabetic retinopathy.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity of detecting moderate non proliferative diabetic retinopathy or more severe DR and/or significant macular edema on a person-specific basis. | Recruitment over 4 months
  If the interval excludes differences of 10% or more (IDx worse than clinical examination), then the IDx system will be considered non-inferior to clinical examination by ophthalmologists. If IDx is non-inferior to clinical examination, a two-sided test of the null hypothesis that the difference in sensitivities is 0 will be conducted to determine if the IDX is superior to clinical examination. 24 McNemar's test for paired proportions will be used to test the difference in proportions.

SECONDARY OUTCOMES:
Specificity (true negatives divided by true negatives plus false positives) at detecting more than moderate non proliferative diabetic retinopathy and/or significant macular edema on a person-specific basis. | Four months
  Secondary Outcome Variables:
  * Specificity on a person-specific basis
  * Sensitivity on an eye-specific basis [Clinical examination only]
  * Specificity on an eye-specific basis [Clinical examination only]
Sensitivity on an eye-specific basis [Clinical examination only] | Four months
  Analysis of secondary outcomes will follow the same approach as for the primary outcome analysis of paired proportions as described above for the comparison of person-specific sensitivity.
Specificity on an eye-specific basis [Clinical examination only] | Four months
  Analysis of secondary outcomes will follow the same approach as for the primary outcome for analysis of paired proportions as described above for the comparison of person-specific sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Graff, MD, Principal Investigator — Barnet Dulaney Perkins Eye Center - Phoenix & Mesa AZ; Brian Privett, MD, Principal Investigator — Iowa Eye Center, Cedar Rapids IA; Timothy Johnson, MD, Principal Investigator — University of Iowa, Iowa City IA; James Major, MD, Principal Investigator — Retina Consultants of Houston - Houston TX (2 locations); Judianne Kellaway, MD, Principal Investigator — Robert Cizik Eye Center - University of Texas Houston
Locations (6):
- United States (6):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Iowa Eye Center, Cedar Rapids, Iowa
  - University of Iowa Department of Ophthalmology and Visual Sciences, Iowa City, Iowa
  - Retina Consultants of Houston, Houston, Texas
  - Robert Cizik Eye Clinic - University of Texas Houston, Houston, Texas